CLINICAL TRIAL: NCT02524262
Title: Slow-release L-cysteine Capsule Prevents Carcinogenic Gastric Acetaldehyde Exposure in Helicobacter-associated Atrophic Gastritis
Brief Title: L-cysteine Prevents Stomach Exposure to Carcinogenic Acetaldehyde
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Per Hellström (Other)
Collaborators: Biohit Oyj, Helsinki, Finland (Unknown); University of Helsinki (Other); Åbo Akademi University (Other); CTC Clinical Trial Consultants AB (Industry)
Responsible Party: Sponsor-Investigator, Per Hellström, Professor, Uppsala University
Organization: Uppsala University (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 620070-SWE-2012
Record Dates: First submitted 2015-08-13; First posted 2015-08-14 (Estimated); Last update posted 2016-01-25 (Estimated); Status verified 2016-01

CONDITIONS: Gastritis, Atrophic
Keywords: atrohpic gastritis; acetaldehyde; ethanol; L-cysteine
MeSH Terms: conditions — Gastritis, Atrophic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Slow-release L-cysteine (Experimental): Oral intake of slow-release L-cysteine 200 mg before challenge with ethanol.
  Interventions: Dietary Supplement: Slow-release L-cysteine
- Placebo (Placebo Comparator): Oral intake of identically-looking placebo capsules
  Interventions: Dietary Supplement: Slow-release L-cysteine

INTERVENTIONS:
Dietary Supplement: Slow-release L-cysteine — Bind and inactivate acetaldehyde formed from ethanol by covalent binding to L-cysteine
  Other Names: Acetium

SUMMARY:
Atrophic gastritis with hypochlorhydric milieu is a risk factor for gastric cancer. Microbes colonizing the acid-free stomach oxidize ethanol into acetaldehyde, a group 1 carcinogen. The aim is to assess gastric production of acetaldehyde and its inert condensation product, non-toxic 4-methyltiazolidine-2-carboxylic acid (MTCA), after alcohol intake under treatment with slow-release L-cysteine or placebo.

Patients with biopsy-confirmed atrophic gastritis, low serum pepsinogen and high gastrin-17 are studied. On separate days, patients will be randomly assigned to receive 200 mg slow-release L-cysteine or placebo, then have intragastric instillation of 15% (0.3 g/kg) ethanol. After intake, gastric concentrations of acetaldehyde, ethanol, L-cysteine and MTCA are analysed for 4 hours.

Expected results show mitigated exposure of the gastric mucosa to acetaldehyde.

DETAILED DESCRIPTION:
Gastric infection with Helicobacter pylori induces chronic active gastritis which over the years develop atrophic gastritis with a hypochlorhydric milieu which is a risk factor for gastric cancer. Microbes colonizing acid-free stomach oxidize ethanol into acetaldehyde, considered a group 1 carcinogen.

The aim of the study is to assess the gastric production of acetaldehyde and its inert condensation product, non-toxic 4-methyltiazolidine-2-carboxylic acid (MTCA), after alcohol intake under treatment with slow-release L-cysteine. Identical placebo tablets will be used for comparison.

Patients with biopsy-confirmed atrophic gastritis, low serum pepsinogen and high gastrin-17 will be studied with case-control design. All subjects will be their own control. On separate days, patients are randomly assigned to receive 200 mg slow-release L-cysteine or placebo, then have intragastric instillation of 15% (0.3 g/kg) ethanol (corresponding to two glasses of wine). After intake, gastric sampling of fluid for a period of four hours is done and concentrations of acetaldehyde, ethanol, L-cysteine and MTCA are analysed.

L-cysteine is expected to decrease gastric acetaldehyde concentrations and increase the MTCA level. Gastric L-cysteine and MTCA concentrations are expected to be maintained over the study period. With placebo, acetaldehyde is expected to be elevated along with ethanol concentrations.

Based on these assumptions slow-release L-cysteine binds acetaldehyde to form inactive MTCA, which remains in gastric juice resulting in reduced local exposure of the gastric mucosa to carcinogenic acetaldehyde.

ELIGIBILITY:
Inclusion Criteria:

* Helicobacter-associated chronic gastritis
* Hypochlorhydria
* Hypergastrinemia
* Hypopepsinogenemia

Exclusion Criteria:

* Active peptic ulcer disease
* Other inflammatory gastrointestinal disease
* Gastrointestinal bleeding
* Gastrointestinal surgery
* Neurological disease
* Alcohol abuse
* Mental disorder
* Not able to sign informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2012-12; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Acetaldehyde concentrations in the stomach | 4 hours
  Binding of acetaldehyde to L-cysteine

SECONDARY OUTCOMES:
4-methyltiazolidine-2-carboxylic acid concentration in the stomach | 4 hours
  Production of inert 4-methyltiazolidine-2-carboxylic acid after binding to L-cysteine

CONTACTS AND LOCATIONS:
Overall Officials: Per M Hellstrom, MD, PhD, Principal Investigator — Uppsala University
Locations (1):
- Uppsala University, Uppsala, Uppsala County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
World J Gastroenterol